CLINICAL TRIAL: NCT02517970
Title: Observing Infant Feeding Interactions
Acronym: MFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Alison Ventura, Assistant Professor, California Polytechnic State University-San Luis Obispo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00001
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Classical Music; Television Show
Keywords: infant feeding; breast-feeding; bottle-feeding; feeding interactions; maternal feeding practices
MeSH Terms: conditions — Breast Feeding; Bottle Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Classical Music versus Television show (Experimental): This is within-subject study; all infants will be exposed to both conditions. Order of presentation will counterbalanced across infants.
  Interventions: Behavioral: Technology distraction

INTERVENTIONS:
Behavioral: Technology distraction — Infants will be fed with classical music playing in the background for one feeding and with a television show playing for the mother to watch during the other.

SUMMARY:
The objective of the proposed research is to conduct a within-subject experimental study that will assess the effect of environmental distractions on a mothers' ability to recognize and feed in response to infants' feeding cues. Investigators hypothesize that mothers will spend significantly more time looking at their technology compared to looking at their infant, which will be negatively associated with the mothers' responsiveness to her infant. This will have a positive association with infant intake during the feeding. Investigators also hypothesize that mothers will show less sensitivity when distracted when compared to when they are not distracted.

ELIGIBILITY:
Inclusion Criteria:

* Mothers must be 18 years or older
* Infants must be between 0-6 months of age

Exclusion Criteria:

* Preterm birth
* Medical conditions that interfere with feeding

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Infant intake within a feeding (mL) | 2-hour period
  Infant intake within a feeding (mL) assessed by weighing the bottle or infant, depending on the type of feeding, before and after the feeding.
Maternal responsiveness | 2-hour period
  Maternal responsiveness to infant cues during a feeding assessed by the Nursing Child Assessment Satellite Training Parent-Child Interaction Feeding Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alison K Ventura, PhD, Principal Investigator — Assistant Professor
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

REFERENCES:
- [Background] Golen RB, Ventura AK. Mindless feeding: Is maternal distraction during bottle-feeding associated with overfeeding? Appetite. 2015 Aug;91:385-92. doi: 10.1016/j.appet.2015.04.078. Epub 2015 May 4. PMID 25953601